CLINICAL TRIAL: NCT02553486
Title: Internationally Adopted Children Quality of Life Study (QUADOP)
Brief Title: Internationally Adopted Children Quality of Life
Acronym: QUADOP
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC15_0062
Record Dates: First submitted 2015-09-15; First posted 2015-09-17 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Children; Quality of Life
Keywords: adoption; children; quality of life

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Internationally adopted children: All internationally adopted children, who arrived in France between 2008 and 2013, living in four French districts
  Interventions: Other: quality of life evaluation

INTERVENTIONS:
Other: quality of life evaluation

SUMMARY:
This study evaluates the global quality of life of foreign born adopted children, one to seven years following their arrival in France. Investigators will assess global health, behavior, school integration for each child who arrived in France between 2008 and 2013, through an online anonymous survey. Investigators, then, will identify variables associated with a lower quality of life in order to improve the support offered to the children.

DETAILED DESCRIPTION:
Investigators will use a known and official quality of life score: the PedsQL®. This score has never been used in this population so investigators will first have to test its internal validity, so that investigators cannot use it in their global evaluation. The second stage will consist of identifying variables associated with a lower quality of life, as previously determined. Investigators will send letters to each family through the adoption department of each area enrolled in our study, to ensure data. Parents and children will be required to login to a safe, anonymous, controlled website in order to input their data. The data will be recorded on the internal server of Nantes University Hospital. This study has been accepted by both the Computing and Liberties Commission (CNIL) and Nantes University Hospital's Ethics group in the field of Health (GNEDS) comities.

ELIGIBILITY:
Inclusion Criteria:

* All international adopted children, who arrived in France between 2008 and 2013, living in four French districts (Loire-Atlantique, Ille et vilaine, Maine et Loire and Finistère) and accepting to fill the on-line questionnaire of the study

Exclusion Criteria:

* Children born in France.
* Children or adoptive parents refusing to participate.

Ages: 1 Month to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All international adopted children, who arrived in France between 2008 and 2013, living in four French districts (Loire-Atlantique, Ille-et-vilaine, Maine et Loire and Finistère)
Sampling Method: Non-Probability Sample
Enrollment: 756 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
International adopted children global quality of life evaluation | up to 9 months
  Global international adopted children quality of life score one to seven years after arrival in France, using a quality of life score : PedsQL®.

SECONDARY OUTCOMES:
Identification of Quality of life low score risk factors | up to 9 months
  Validation of the questionnaire in our population; Highlight the determiners of a bad quality of life (after dichotomization of the population, investigators will compare participants who have a score under one standard deviation to those who have a better score).

REFERENCES:
- [Background] Upton P, Eiser C, Cheung I, Hutchings HA, Jenney M, Maddocks A, Russell IT, Williams JG. Measurement properties of the UK-English version of the Pediatric Quality of Life Inventory 4.0 (PedsQL) generic core scales. Health Qual Life Outcomes. 2005 Apr 1;3:22. doi: 10.1186/1477-7525-3-22. PMID 15804349
- [Background] Hjern A, Lindblad F, Vinnerljung B. Suicide, psychiatric illness, and social maladjustment in intercountry adoptees in Sweden: a cohort study. Lancet. 2002 Aug 10;360(9331):443-8. doi: 10.1016/S0140-6736(02)09674-5. PMID 12241716
- [Background] de Monleon JV, Huet F. [Usefulness of management of adopted children born in foreign countries]. Arch Pediatr. 2000 Oct;7(10):1039-40. doi: 10.1016/s0929-693x(00)00310-9. No abstract available. French. PMID 11075257